CLINICAL TRIAL: NCT01721109
Title: A Phase 2/3, Open-Label Study of the Pharmacokinetics, Safety, and Antiviral Activity of the Elvitegravir/ Cobicistat/Emtricitabine/Tenofovir Disoproxil Fumarate Single Tablet Regimen (STR) in HIV-1 Infected Antiretroviral Treatment-Naive Adolescents
Brief Title: Pharmacokinetics, Safety, and Efficacy of Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Disoproxil Fumarate Single Tablet Regimen (STR) in Adolescents
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-236-0112; 2015-000313-40 (EudraCT Number)
Record Dates: First submitted 2012-11-01; First posted 2012-11-05 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-07

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV Infections
Keywords: Adolescents; HIV-1; HIV; Treatment Naive
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EVG/COBI/FTC/TDF (Experimental): Participants will receive treatment for 48 weeks and then had the option to enter an Extension Phase to receive EVG/COBI/FTC/TDF until 1) the age of 18, 2) EVG/COBI/FTC/TDF becomes commercially available in the country the participant is enrolled, or 3) Gilead elects to terminate the development of EVG/COBI/FTC/TDF in that country.
  Interventions: Drug: EVG/COBI/FTC/TDF

INTERVENTIONS:
Drug: EVG/COBI/FTC/TDF — 150/150/200/300 mg STR administered orally once daily with food
  Other Names: Stribild®

SUMMARY:
The primary objectives of this study are to evaluate the steady-state pharmacokinetics (PK) and confirm the dose of the elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate (EVG/COBI/FTC/TDF) single-tablet regimen (STR) (Part A) and to evaluate the safety and tolerability of EVG/COBI/FTC/TDF STR through Week 48 (Part B) in HIV-1 infected, antiretroviral (ARV) treatment-naive adolescents.

A total of 50 adolescent participants (12 to < 18 years of age) will be enrolled to receive EVG/COBI/FTC/TDF as follows:

* Part A: Twelve to 16 eligible participants will be enrolled to evaluate steady-state PK, and confirm the dose, with the intent to enroll at least 4 participants 12 to < 15 and at least 4 participants 15 to < 18 years of age.
* Part B: Following confirmation of EVG exposure in at least 12 participants from Part A, 34 to 38 participants in addition to those enrolled in Part A will be enrolled to evaluate the safety, tolerability, and antiviral activity of EVG/COBI/FTC/TDF STR.

ELIGIBILITY:
Key Inclusion Criteria:

* 12 years to < 18 years of age at baseline
* Able to give written assent prior to any screening evaluations
* Parent or guardian able to give written informed consent prior to any screening evaluations and willing to comply with study requirements
* Plasma HIV-1 RNA levels of ≥ 1,000 copies/mL
* CD4+ cell count > 100 cells/µL
* Weight ≥ 35 kg (77 lbs)
* Screening genotype report must show sensitivity to FTC and TDF
* Able to swallow oral tablets
* Adequate renal function
* Clinically normal ECG
* Documented screening for active pulmonary tuberculosis per local standard of care within 6 months of a screening visit
* Hepatic transaminases ≤ 5 x upper limit of normal
* Total bilirubin ≤ 1.5 mg/dL, or normal direct bilirubin
* Individuals with a positive Hepatitis B surface antigen screening test can participate in the study, providing that alternate therapy (other than TDF) for chronic Hepatitis B infection is available as a part of local standard of care
* Adequate hematologic function
* Negative serum pregnancy test for all females
* Males and females of childbearing potential must agree to utilize highly effective contraception methods while on study treatment or agree to abstain from heterosexual intercourse throughout the study period and for 30 days following the last dose of study drug
* Males must agree to utilize a highly effective method of contraception during heterosexual intercourse throughout the study period and for 30 days following discontinuation of investigational medicinal product
* Must be willing and able to comply with all study requirements
* Life expectancy ≥ 1 year

Key Exclusion Criteria:

* A new AIDS-defining condition diagnosed within the 30 days prior to screening
* Prior treatment with any approved or investigational or experimental anti HIV-1 drug for any length of time (other than that given for prevention of mother-to-child transmission)
* Evidence of active pulmonary or extra-pulmonary tuberculosis disease within 3 months of the screening visit
* Anticipated to require rifamycin treatment for mycobacterial infection while participating in the study. Note: prophylactic Isoniazid (INH) therapy for latent tuberculosis (TB) treatment is allowed.
* Individuals experiencing decompensated cirrhosis
* Pregnant or lactating females
* Have any serious or active medical or psychiatric illness which would interfere with treatment, assessment, or compliance with the protocol. This would include uncontrolled renal, cardiac, hematological, hepatic, pulmonary, endocrine, central nervous, gastrointestinal, vascular, metabolic, immunodeficiency disorders, active infection, or malignancy that are clinically significant or requiring treatment within 30 days prior to the study dosing.
* Current alcohol or substance abuse that will potentially interfere with compliance
* Have history of significant drug sensitivity or drug allergy
* Known hypersensitivity to the study drugs, the metabolites or formulation excipients
* Have been treated with immunosuppressant therapies or chemotherapeutic agents within 3 months of study screening or expected to receive these agents during the study
* A history of malignancy within the past 5 years or ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous carcinoma
* Have previously participated in an investigational trial involving administration of any investigational agent within 30 days prior to the study dosing
* Participation in any other clinical trial without prior approval from sponsor is prohibited while participating in this trial
* Receiving ongoing therapy with any disallowed medications, including drugs not to be used with EVG, COBI, FTC, TDF or individuals with any known allergies to the excipients of EVG/COBI/FTC/TDF STR tablets

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2012-12-06 (Actual); Primary Completion 2015-10-22 (Actual); Study Completion 2018-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (18):
- United States (7):
  - East Bay AIDS Center Medical Group, Oakland, California
  - University of South Florida - Department of Pediatrics, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - New York University School of Medicine, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
- South Africa (7):
  - Rahima Moosa Mother and Child Hospital (Wits), Johannesburg, Gauteng
  - Dr Latiff Private Practice, Durban, KwaZulu-Natal
  - Desmond Tutu HIV Research Centre, Cape Town
  - Mpati Medical Center, Dundee
  - Clinical HIV Research Unit, Johannesburg
  - Perinatal HIV Research Unit, Soweto
  - University of Stellenbosch, Stellenbosch
- Thailand (4):
  - The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT), Bangkok
  - Siriraj Hospital, Mahidol University, Bangkok
  - Queen Savang Vadhana Memorial Hospital, Chon Buri
  - Srinakarind Hospital, Khon Kaen

REFERENCES:
- [Result] Gaur A, Fourie J, Chokephaibulkit K, Bekker L-G, Yin X, Custodio J, Bennett S, Cheng A, Quirk E. Pharmacokinetics, Efficacy and Safety of an Integrase Inhibitor-Based Single-Tablet Regimen in HIV-Infected Treatment-Naïve Adolescents. 21st Conference on Retroviruses and Opportunistic Infections (CROI). March 2014. Boston, MA, USA
- [Result] Chokephaibulkit K, Gaur A, Fourie J, Bekker L-G, Shao Y, Custodio J, Bennett S, Cheng A, Quirk E. Safety and Efficacy of the Integrase Inhibitor-Based Stribild Single-Tablet Regimen in HIV-Infected Adolescents Through 24 Weeks of Treatment. 20th International AIDS Conference. July 2014. Melbourne, Australia
- [Result] Porter DP, Bennett S, Quirk E, Miller MD, White KL. Lack of Emergent Resistance in HIV-1-Infected Adolescents on Elvitegravir-Based STRs. 22nd Conference on Retroviruses and Opportunistic Infections (CROI). February 2015. Seattle, WA, USA
- [Result] Kizito H, Gaur A, Prasitsuebsai W, Rakhmanina N, Chokephaibulkit K, Fourie J, Bekker LG, Shao Y, Bennett S, Quirk E. Changes in renal laboratory markers and bone mineral density in treatment-naïve HIV-1-infected adolescents initiating INSTI-based single-tablet regimens containing tenofovir alafenamide (TAF) or tenofovir disoproxil fumarate (TDF). 8th IAS Conference on HIV Pathogenesis, Treatment & Prevention. July 2015. Vancouver, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, South Africa, and Thailand. The first participant was screened on 06 December 2012. The last study visit occurred on 29 January 2018.
Pre-assignment Details: 56 participants were screened.
Groups:
- EVG/COBI/FTC/TDF: Elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate (EVG/COBI/FTC/TDF) (150/150/200/300 mg) single-tablet regimen (STR) administered orally once daily with food for 48 weeks, followed by EVG/COBI/FTC/TDF (150/150/200/300 mg) during the optional extension phase.
Period: Overall Study
Arm/Group | EVG/COBI/FTC/TDF
Started | 50
Completed | 43 (34 participants transitioned to commercial Stribild or to an individual patient use (IPU) program)
Not Completed | 7
Not completed — Lack of Efficacy | 1
Not completed — Non- Compliance with Study Drug | 3
Not completed — Withdrew Consent | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all participants who received at least 1 dose of study drug.
Groups:
- EVG/COBI/FTC/TDF: EVG/COBI/FTC/TDF (150/150/200/300 mg) STR administered orally once daily with food for 48 weeks, followed by EVG/COBI/FTC/TDF (150/150/200/300 mg) during the optional extension phase
Arm/Group | EVG/COBI/FTC/TDF
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 15 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 14
  Black | 34
  White | 1
  Other | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 47
  Not Permitted | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14
  South Africa | 22
  Thailand | 14
HIV-1 RNA [Mean (Standard Deviation); unit: log10 copies/mL] | 4.60 (0.551)
HIV-1 RNA Category [Count of Participants; unit: Participants]
  ≤ 100,000 copies/mL | 40
  > 100,000 copies/mL | 10
CD4 Cell Count [Mean (Standard Deviation); unit: cells/µL] | 399 (127.6)
CD4 Cell Count Category [Count of Participants; unit: Participants]
  ≤ 199 cells/µL | 2
  200 ≥ and ≤ 349 cells/µL | 16
  350 ≥ and ≤ 499 cells/µL | 22
  ≥ 500 cells/µL | 10

OUTCOME MEASURES:

1. Primary Outcome: For Part A, Pharmacokinetic (PK) Parameter: AUCtau of EVG
Description: AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
Time Frame: Predose, 2, 4, 4.5, 5, 8, and 12 hours postdose on Day 10
Population: PK Substudy Analysis Set: all enrolled and treated participants from Part A who had evaluable steady-state pharmacokinetic profiles of the respective analyte of interest at the Day 10 intensive PK visit.
Measure: Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | EVG/COBI/FTC/TDF
Number analyzed (Participants) | 14
ng•h/mL | 31620.9 (13978.07)
Statistical Analysis 1: Comparison: EVG/COBI/FTC/TDF; Test type: Equivalence — A sample size of 14 participants was estimated to provide over 95% power to show pharmacokinetic equivalence between adult and adolescent participants. EVG population PK from historical adult data was used for comparison. The inter-subject standard deviation (natural log scale) of EVG AUCtau observed in the population PK data was 0.31 (historical data); Geometric least squares mean ratio = 1.3029, 90% CI 2-sided [1.0479 to 1.6200]

2. Primary Outcome: Incidence of Treatment-Emergent Serious Adverse Events (SAEs) and All Treatment-Emergent Adverse Events (AEs)
Time Frame: Up to Week 48 plus 30 days
Population: Safety Analysis Set: all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | EVG/COBI/FTC/TDF
Number analyzed (Participants) | 50
Participants
  SAEs | 4
  AEs | 45

3. Secondary Outcome: For Part A, PK Parameter: Ctau of EVG, FTC, Tenofovir (TFV), and COBI
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval.
Time Frame: Predose, 2, 4, 4.5, 5, 8, and 12 hours postdose on Day 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | EVG/COBI/FTC/TDF
Number analyzed (Participants) | 14
ng/mL
  EVG | 579.3 (455.20)
  FTC | 102.6 (30.85)
  TFV | 86.6 (23.58)
  COBI | 39.7 (68.52)

4. Secondary Outcome: For Part A, PK Parameter: Cmax of EVG, FTC, TFV, and COBI
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: Predose, 2, 4, 4.5, 5, 8, and 12 hours postdose on Day 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | EVG/COBI/FTC/TDF
Number analyzed (Participants) | 14
ng/mL
  EVG | 2624.3 (1239.64)
  FTC | 2217.4 (664.64)
  TFV | 438.5 (170.69)
  COBI | 1500.4 (975.29)

5. Secondary Outcome: For Part A, PK Parameter: AUCtau of FTC, TFV, and COBI
Description: as for outcome 1
Time Frame: Predose, 2, 4, 4.5, 5, 8, and 12 hours postdose on Day 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | EVG/COBI/FTC/TDF
Number analyzed (Participants) | 14
ng•h/mL
  FTC | 15136.5 (4702.06)
  TFV | 4450.7 (1312.27)
  COBI | 11884.8 (11220.94)

6. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Weeks 24 and 48 as Defined by the FDA Snapshot Analysis
Time Frame: Weeks 24 and 48
Population: Full Analysis Set: all participants who were enrolled in the study and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | EVG/COBI/FTC/TDF
Number analyzed (Participants) | 50
percentage of participants
  Week 24 | 88.0
  Week 48 | 88.0

7. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 400 Copies/mL at Weeks 24 and 48 as Defined by the FDA Snapshot Analysis
Time Frame: Weeks 24 and 48
Population: Full Analysis Set: all participants who were enrolled in the study and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | EVG/COBI/FTC/TDF
Number analyzed (Participants) | 50
percentage of participants
  Week 24 | 94.0
  Week 48 | 92.0

8. Secondary Outcome: Change From Baseline in Plasma log10 HIV-1 RNA at Weeks 24 and 48
Time Frame: Baseline; Weeks 24 and 48
Population: Full Analysis Set: all participants who were enrolled in the study and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | EVG/COBI/FTC/TDF
Number analyzed (Participants) | 50
log10 copies/mL
  Change at Week 24 | -3.08 (0.922)
  Change at Week 48 | -3.16 (0.705)

9. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Weeks 24 and 48
Time Frame: Baseline; Weeks 24 and 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | EVG/COBI/FTC/TDF
Number analyzed (Participants) | 49
cells/µL
  Change at Week 24 | 178 (165.4)
  Change at Week 48: number analyzed (Participants) | 48
  Change at Week 48 | 229 (245.3)

10. Secondary Outcome: Change From Baseline in CD4 Percentage at Weeks 24 and 48
Time Frame: Baseline; Weeks 24 and 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | EVG/COBI/FTC/TDF
Number analyzed (Participants) | 49
percentage
  Change at Week 24 | 7.4 (4.70)
  Change at Week 48: number analyzed (Participants) | 48
  Change at Week 48 | 8.1 (5.34)

ADVERSE EVENTS:
Time Frame: Baseline up to the last dose date plus 30 days (maximum exposure: 250.7 weeks)
Description: Safety Analysis Set: all participants who received at least 1 dose of study drug.
Arm/Group | EVG/COBI/FTC/TDF
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 5/50
Other Adverse Events (participants affected / at risk) | 46/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EVG/COBI/FTC/TDF (N=50)
Anaemia (Blood and lymphatic system disorders) | 1
Food poisoning (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Immune reconstitution inflammatory syndrome (Immune system disorders) | 1
Disseminated tuberculosis (Infections and infestations) | 1
Gastroenteritis shigella (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Suicidal behaviour (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EVG/COBI/FTC/TDF (N=50)
Diarrhoea (Gastrointestinal disorders) | 8
Haemorrhoids (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 8
Toothache (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 10
Pyrexia (General disorders) | 3
Bronchitis (Infections and infestations) | 4
Influenza (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 4
Oral herpes (Infections and infestations) | 3
Oropharyngeal gonococcal infection (Infections and infestations) | 3
Pharyngitis (Infections and infestations) | 6
Proctitis gonococcal (Infections and infestations) | 3
Respiratory tract infection viral (Infections and infestations) | 3
Secondary syphilis (Infections and infestations) | 3
Tonsillitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 18
Urinary tract infection (Infections and infestations) | 3
Skin abrasion (Injury, poisoning and procedural complications) | 3
Weight decreased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 3
Vitamin D deficiency (Metabolism and nutrition disorders) | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 12
Acne (Skin and subcutaneous tissue disorders) | 8
Dermatitis (Skin and subcutaneous tissue disorders) | 3
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years